CLINICAL TRIAL: NCT03027388
Title: Phase II Trial of LB100, a Protein Phosphatase 2A Inhibitor, in Recurrent Glioblastoma
Brief Title: Protein Phosphatase 2A Inhibitor, in Recurrent Glioblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Eric Burton, Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 170037; 17-C-0037
Record Dates: First submitted 2017-01-18; First posted 2017-01-23 (Estimated); Results first posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Astrocytoma, Grades II, III and IV; Glioblastoma Multiforme; Giant Cell Glioblastoma; Glioma; Oligodendrogliomas
Keywords: Brain Tumor; Blood Brain Barrier; Pharmacokinetics; Pharmacodynamics
MeSH Terms: conditions — Astrocytoma; Glioblastoma; Glioma; Oligodendroglioma; Brain Neoplasms | interventions — LB100

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1/LB100 Protein Phosphatase 2A Inhibitor, in Recurrent Glioblastoma (Experimental): Treatment with LB100
  Interventions: Drug: LB-100

INTERVENTIONS:
Drug: LB-100 — LB-100 will be infused over 2 hours via intravenous (IV) infusion 2 to 4 hours before surgery. The dose established from a Phase I study will be 2.33 mg/m^2.

SUMMARY:
Background:

The brain is separated from the rest of the blood stream by the blood-brain barrier. This is like a filter that protects the brain. But is also a challenge when medicines need to get into the brain. Researchers want to give the new drug LB100 to people before brain tumor surgery. They will measure how much LB100 is in the blood and how much gets into the brain. This may help with the use of LB100 to treat brain tumors in the future.

Objective:

To see if LB100 can pass into the brain.

Eligibility:

People at least 18 years old with a brain tumor that requires surgery.

Design:

Participants will be screened with:

Physical exam

Medical history

Blood tests

Neurosurgery evaluation

Scans

Heart tests

Tumor sample. This can be from a previous procedure.

Participants will have their brain surgery at the Clinical Center.

Participants will get a dose of the study drug through a plastic tube in a vein for 2 hours during surgery.

Participants will have blood taken 7 times in the 8 hours after getting the study drug.

Tumor samples will be taken during surgery.

Participants will have a heart test after getting the study drug. Sticky pads on the skin will measure electrical activity of the heart.

Two-three weeks after leaving the hospital, participants will have a follow-up visit. They will have a physical exam and blood tests.

One month after surgery, they will be contacted in person or by phone to see how they are doing.

DETAILED DESCRIPTION:
Background:

* Primary gliomas are an incurable disease in spite of aggressive multimodality therapy consisting of craniotomy, irradiation, and chemotherapy. Therapeutic options for patients with recurrent glioma are limited, and there is an unmet need to identify more effective agents.
* LB100, a water-soluble small molecule novel protein phosphatase 2A (PP2A) inhibitor, was commercially developed through a Cooperative Research and Development Agreement (CRADA) based on our previous intramural research. This compound has shown to be effective in a variety of cancer types in both in vitro and in vivo models. Preclinical studies indicate LB100 has in vitro and in vivo activity as a single agent as well as potentiating the effect of cytotoxic agents including temozolomide, docetaxel, doxorubicin, and ionizing radiation. LB100 is active in combination with temozolomide or doxorubicin against xenografts of glioblastoma, neuroblastoma, pheochromocytoma, breast cancer, fibrosarcoma, and melanoma.
* A complete phase I study of LB100 has established its safety and the recommended phase II dose (2.33 mg/m^2, daily for three days every 3 weeks).
* Although it is a polar compound, rodent studies suggest LB100 has activity in the brain.
* Whether LB100 can across the human blood brain barrier (BBB), and at what concentration relative to the plasma level is not known. Characterizing these parameters is important because:

  * 1) Our ongoing in vitro studies indicate that LB100 has distinct mechanisms of action at different drug concentrations (e.g., nM versus uM);
  * 2) There are other brain tumors lacking effective medical therapies but without a BBB. Characterizing the LB100 BBB penetration profile will assist in defining its optimal clinical indication.

Objective:

-To determine the pharmacokinetic (PK) properties of LB100 in glioma tumor tissues.

Eligibility:

* Patients with histologically proven glioblastoma and grades II-III astrocytomas and oligodendrogliomas.
* A clear clinical indication for another surgical resection must be present.
* Subjects must be greater than or equal to 18 years old.
* Karnofsky performance status of greater than or equal to 60%.
* Patients must have adequate organ function.

Design:

* This is a two stage Phase II, open label, single institution study to determine the PK and pharmacodynamic (PD) profile of LB100.
* The dose (established from a Phase I study) will be 2.33 mg/m^2 delivered intravenously over 2 hours.
* PK and PD effect of LB100 treated tissues will only be evaluated with pathologic confirmation of recurrent tumor. Resected material demonstrating chemoradiation treatment effect or inflammatory response will not be included in the analysis.
* PK will be determined by quantitating LB100 in tumor tissues removed at various time points.
* The primary endpoint is PK response, defined as a binary variable indicating the presence/absence of LB100 in tumor tissues.
* PD effect is defined as statistically significant elevation of phospho-proteins in treated tumor tissues compared to untreated glioma specimens. Untreated inter-patient baseline variance and standard deviation (SD) will be calculated. Post-treatment PD effect difference greater than 2.5 times the baseline SD is statistically significant at the .05 significance level. Due to relatively small sample size, t-distribution is to be used to calculate the cutoff defining the PD response.
* Up to 25 patients may be enrolled to obtain 8 evaluable subjects. A two-stage design will be used. Five patients will be initially treated. If at least one of five demonstrates PK activity, 3 additional subjects will be enrolled. PK effect will be declared to be significant if at least 2 of the 8 patients demonstrate a PK response (presence of LB100 in tumor tissue).

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have histologically confirmed glioblastoma/gliosarcoma, grades II-III astrocytoma and oligodendroglioma.
* Patients must have recurrent disease for which there is a clinical indication for resection.
* Age greater than or equal to18 years.
* Karnofsky greater than or equal to 60%.
* Patients must have adequate bone marrow function (white blood count (WBC) greater than or equal to 3,000/uL absolute neutrophil count (ANC) greater than or equal to 1,500/mm^3, platelet count of greater than or equal to 100,000/mm^3, and hemoglobin greater than or equal to 10 gm/dL), adequate liver function (SGOT and bilirubin < 2 times upper limit of normal (ULN). These tests must be performed within 28 days prior to receiving drug. Eligibility level for hemoglobin may be reached by transfusion.
* Patients must have a serum creatinine of <=1.7 mg/dL. If the serum creatinine is greater than 1.7 mg/dl, a 24-hour urine creatinine clearance will be obtained and if the result of this study is within normal limits*, the patient would be eligible to enroll onto study. This test must be performed within 28 days prior to registrationreceiving drug. (*Normal Creatinine Clearance Range: Male: 90 - 130 ml/min; Female: 80 - 125 ml/min)
* Patients must be in adequate general medical health to safely tolerate a craniotomy.
* At the time of registration, all subjects must be removed greater than or equal to 28 days from any investigational agents.
* The effects of LB100 on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Ability of subject to understand and the willingness to sign a written informed consent document indicating that they are aware of the investigational nature of this study, and that this is not a therapeutic clinical trial.

EXCLUSION CRITERIA:

* Patients who are receiving any other investigational agents.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients unwilling to undergo craniotomy.
* Pregnant women are excluded from this study because the safety of Protein Phosphatase 2A (PP2A) inhibition on a developing fetus has not been established. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with LB100, breastfeeding should be discontinued if the mother is treated with LB100.
* Patients may not have had prior chemotherapy or biologic therapy in the 4 weeks prior to study entry. For patients who have been treated with targeted therapy, 5 half-lives of that therapy (or 28 days, whichever is shorter) must have passed prior to enrollment in the study.
* Known human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with LB100. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.
* Patients who are receiving strong cytochromes P450 (CYP450) inducers or inhibitors are ineligible
* Recruitment Strategies

Patients with recurrent disease will be identified by the Neuro-Oncology Branch, Clinical Center. This study will be posted on National Institutes of Health (NIH) websites and on NIH Social media forums.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-01-09 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric C Burton, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI).

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2017-C-0037.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 1/LB100 Protein Phosphatase 2A Inhibitor, in Recurrent Glioblastoma
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 1/LB100 Protein Phosphatase 2A Inhibitor, in Recurrent Glioblastoma
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.17 (7.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With the Presence of Drug in the Tumor Tissue
Description: Participants tumor tissue was examined to determine the presence of drug in the tumor tissue.
Time Frame: an average of 5.5 hours after drug administration
Population: 2/7 were not analyzed because no tumor was found on analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | 1/LB100 Protein Phosphatase 2A Inhibitor, in Recurrent Glioblastoma
Number analyzed (Participants) | 5
Participants | 2

2. Secondary Outcome: Plasma Concentration and Calculated LB100
Description: Blood samples for the determination of plasma levels of LB-100 will be obtained from each participant. Plasma concentrations of LB100 will be determined at each time point. LC-MS-MS assay that can measure LB-100 in human plasma. Assay range is 2.0 -1000 ng/mL. A higher value is better because it would have made it more likely drug could penetrate the blood brain barrier at therapeutic levels.
Time Frame: Pre-dose; End of infusion (2 hours post-start); 30 minutes post LB100 infusion completion; 1 hour post LB-100 infusion completion; 2 hours post LB100 infusion completion; 4 hours post LB100 infusion completion; 8 hours post LB100 infusion completion
Measure: Median (Full Range); unit: (rounded)nM
Arm/Group | 1/LB100 Protein Phosphatase 2A Inhibitor, in Recurrent Glioblastoma
Number analyzed (Participants) | 5
(rounded)nM
  Pre-dose | 0.0 [0 to 0]
  End of infusion (2 hours post-start) | 575 [354 to 772]
  30 minutes post LB100 infusion completion | 534 [291 to 626]
  1 hour post LB-100 infusion completion | 355 [251 to 633]
  2 hours post LB100 infusion completion | 192 [174 to 263]
  4 hours post LB100 infusion completion | 80 [30 to 150]
  8 hours post LB100 infusion completion | 16 [07 to 71]

3. Secondary Outcome: Concentration of LB100
Description: Concentration of LB100 in glioma tumor tissue when a known non-toxic dose of LB100 is delivered intravenously. Glioma tissue sampling to detect and quantify LB100 will be performed by assaying phospho-protein expression in glioma tissue resected prior to and after infusion of LB100. These are values for the LB100 in the tumor which was done at one timepoint.
Time Frame: average of 5.5 hours after infusion
Measure: Median (Full Range); unit: nM
Arm/Group | 1/LB100 Protein Phosphatase 2A Inhibitor, in Recurrent Glioblastoma
Number analyzed (Participants) | 5
nM | 0.18 [0 to 0.67]

4. Secondary Outcome: Changes in Phospho-protein Expression in Circulating Peripheral Blood Mononuclear Cells (PBMC)
Description: Changes in phospho-protein expression in circulating PBMC. Pharmacodynamic (PD) response is defined as statistically significant elevation of phospho-protein expression in treated tumor tissues compared to untreated glioma specimens. Post-treatment PD effect (as measured by increase in tumor tissue phospho-protein expression) difference greater than 2.5 times the baseline standard deviation (SD) is statistically significant at the .05 significance level.
Time Frame: as for outcome 2
Population: Data was not collected.
Arm/Group | 1/LB100 Protein Phosphatase 2A Inhibitor, in Recurrent Glioblastoma
Number analyzed (Participants) | 0

5. Secondary Outcome: Maximum Observed Plasma Concentration of LB100 (Cmax)
Description: The maximum observed analyte concentration in serum was reported.
Time Frame: as for outcome 2
Measure: Median (Full Range); unit: ng/mL
Arm/Group | 1/LB100 Protein Phosphatase 2A Inhibitor, in Recurrent Glioblastoma
Number analyzed (Participants) | 5
ng/mL | 156 [95 to 207]

6. Secondary Outcome: Area Under the Plasma Concentration vs. Time Curve Extrapolated to Infinity (AUC(INF)
Description: AUC is a measure of the serum concentration of LMB100 over time. It is used to characterize drug absorption.
Time Frame: as for outcome 2
Measure: Median (Full Range); unit: hr*ng/mL
Arm/Group | 1/LB100 Protein Phosphatase 2A Inhibitor, in Recurrent Glioblastoma
Number analyzed (Participants) | 5
hr*ng/mL | 438 [319 to 585]

7. Secondary Outcome: Plasma Half-Life of Drug LB100
Description: Plasma decay half-life is the time measured for the plasma concentration of the drug to decrease by one half.
Time Frame: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | 1/LB100 Protein Phosphatase 2A Inhibitor, in Recurrent Glioblastoma
Number analyzed (Participants) | 5
Hours | 1.20 [1.09 to 1.46]

8. Secondary Outcome: Time to Maximum Observed Plasma Concentration of LMB100 (Tmax)
Description: Time to maximum observed plasma concentration of LMB100 (Tmax).
Time Frame: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | 1/LB100 Protein Phosphatase 2A Inhibitor, in Recurrent Glioblastoma
Number analyzed (Participants) | 5
Hours | 2.10 [2.0 to 2.63]

9. Secondary Outcome: Total Clearance (CL) of LMB100
Description: The CL is a quantitative measure of the rate at which a drug substance is removed from the body.
Time Frame: as for outcome 2
Measure: Median (Full Range); unit: L/hr
Arm/Group | 1/LB100 Protein Phosphatase 2A Inhibitor, in Recurrent Glioblastoma
Number analyzed (Participants) | 5
L/hr | 10.4 [7.13 to 14.7]

10. Secondary Outcome: Volume of Distribution (Vd) of LMB100
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug.
Time Frame: as for outcome 2
Measure: Median (Full Range); unit: L
Arm/Group | 1/LB100 Protein Phosphatase 2A Inhibitor, in Recurrent Glioblastoma
Number analyzed (Participants) | 5
L | 20.1 [12.2 to 31.3]

11. Secondary Outcome: Brain Concentration
Description: Drug amount in brain as a percent of drug in plasma.
Time Frame: as for outcome 2
Measure: Median (Full Range); unit: percent
Arm/Group | 1/LB100 Protein Phosphatase 2A Inhibitor, in Recurrent Glioblastoma
Number analyzed (Participants) | 5
percent | 0.30 [0.0 to 0.45]

12. Secondary Outcome: Brain Penetration
Description: Concentration of drug in brain tumor tissue. Brain penetration is measured as "drug amount in a brain as a percent of drug in plasma.
Time Frame: as for outcome 2
Measure: Median (Full Range); unit: Percent
Arm/Group | 1/LB100 Protein Phosphatase 2A Inhibitor, in Recurrent Glioblastoma
Number analyzed (Participants) | 5
Percent | 0.26 [0 to 0.7]

13. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 39 months and 6 days.
Measure: Count of Participants; unit: Participants
Arm/Group | 1/LB100 Protein Phosphatase 2A Inhibitor, in Recurrent Glioblastoma
Number analyzed (Participants) | 7
Participants | 7

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 39 months and 6 days.
Arm/Group | 1/LB100 Protein Phosphatase 2A Inhibitor, in Recurrent Glioblastoma
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 1/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1/LB100 Protein Phosphatase 2A Inhibitor, in Recurrent Glioblastoma (N=7)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1/LB100 Protein Phosphatase 2A Inhibitor, in Recurrent Glioblastoma (N=7)
Agitation (Psychiatric disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Dysphasia (Nervous system disorders) | 1 (1)
Ear and labyrinth disorders - Other, impacted cerumen (Ear and labyrinth disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Facial muscle weakness (Nervous system disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 5 (7)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (3)
Muscle weakness left-sided (Nervous system disorders) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Skin induration (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-06-02): https://cdn.clinicaltrials.gov/large-docs/88/NCT03027388/Prot_SAP_000.pdf
  • Informed Consent Form (2022-07-13): https://cdn.clinicaltrials.gov/large-docs/88/NCT03027388/ICF_001.pdf